CLINICAL TRIAL: NCT01494584
Title: Open-label, Multiple Dose Study to Evaluate the Parmacokinetics, Safety and Tolerability of Ezogabine/Retigabine as Adjunctive Treatment in Subjects Aged From 12 Years to Less Than 18 Years With Partial Onset Seizures or Lennox-Gastaut Syndrome
Brief Title: Study in Pediatric Subjects With Epilepsy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated after placing the study on hold at the request of the FDA
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113284
Record Dates: First submitted 2011-12-01; First posted 2011-12-19 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ezogabine/retigabine (Experimental): ezogabine dose escalation
  Interventions: Drug: ezogabine/retigabine

INTERVENTIONS:
Drug: ezogabine/retigabine — ezogabine dose escalation

SUMMARY:
This is an open-label study to evaluate the pharmacokinetics, safety and tolerability of ezogabine/retigabine in subjects aged 12 years to less than 18 years with uncontrolled partial onset seizures or Lennos-Gastaut syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Between 12 and 18 years of age.
* Diagnosis of uncontrolled partial onset seizures (with or without secondarily generalized seizures) or Lennox-Gastaut syndrome.
* Taking between one and three antiepileptic drugs.
* Able to swallow tablets.
* Females must be of : (1) Non-childbearing potential or (2) Child-bearing potential and agrees to use acceptable contraception.

Exclusion Criteria:

* Epilepsy secondary to progressive cerebral disease, tumor or any progressive neurodegenerative disease.
* History of status epilepticus in the last six months.
* Currently treated with felbamate or has been treated with vigabatrin within the past 6 months.
* Following the ketogenic diet.
* Suicidal intent or history of suicide attempt in the last 2 years.
* Elevated liver enzymes or abnormal kidney function.
* Current disturbance of micturition or known urinary obstructions.
* History of vesicoureteric reflux.
* Abnormal post-void residual bladder ultrasound.
* Urinary retention and/or required urinary catheterization in the preceding 6 months.
* Abnormal urine sample at screening/.baseline.
* Abnormal blood sample at screening.
* Clinically significant arrhythmias.
* Abnormal ECG at screening.
* BMI lower than the 10th percentile for age and gender or subject weighs less than 30kg.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2012-07-25 (Actual); Primary Completion 2013-04-29 (Actual); Study Completion 2013-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Wellington, Florida
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Dallas, Texas

REFERENCES:
- [Background] Tompson DJ, Buraglio M, Andrews SM, Wheless JW. Adolescent Clinical Development of Ezogabine/Retigabine as Adjunctive Therapy for Partial-Onset Seizures: Pharmacokinetics and Tolerability. J Pediatr Pharmacol Ther. 2016 Sep-Oct;21(5):404-412. doi: 10.5863/1551-6776-21.5.404. PMID 27877093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolled participants (par.) were aged 12 years to less than 18 years with partial onset seizures or Lennox-Gastaut syndrome (LGS), and were required to be on at least 1 but not more than 3 anti-epileptic therapies without achieving complete control of their seizures.
Pre-assignment Details: A total of 5 par. who met the eligibility criteria were assigned to Regimen A (>50 kilograms [kg]) or B (30 to <=50 kg) based on body weight and entered a 2-week Screening phase, followed by a dosing phase (up to 5 weeks). Upon completion of the dosing phase, par. either entered a follow-up phase or a separate extension study.
Groups:
- Ezogabine/Retigabine: Participants recieved an initial dose of ezogabine/retigabine 300 milligrams (mg) per day administered as 100 mg immediate release (IR) tablets three times a day (TID) orally and underwent weekly up-titration at Weeks 1, 3, and 5. Dose titration occurred no more than once per week, with participants receiving up-titrated daily doses of 450 mg (150 mg TID), 600 mg (200 mg TID), 750 mg (250 mg TID), and 900 mg (300 mg TID) at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
Period: Overall Study
Arm/Group | Ezogabine/Retigabine
Started | 5
Completed | 4
Not Completed | 1
Not completed — Study Closed/Terminated | 1

BASELINE CHARACTERISTICS:
Groups:
- Ezogabine/Retigabine: Participants received an initial dose of ezogabine/retigabine 300 milligrams (mg) per day administered as 100 mg immediate release (IR) tablets three times a day (TID) orally and underwent weekly up-titration at Weeks 1, 3, and 5. Dose titration occurred no more than once per week, with participants receiving up-titrated daily doses of 450 mg (150 mg TID), 600 mg (200 mg TID), 750 mg (250 mg TID), and 900 mg (300 mg TID) at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
Arm/Group | Ezogabine/Retigabine
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.6 (1.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  White-White/Caucasian/European Heritage | 5

OUTCOME MEASURES:

1. Primary Outcome: The Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUC[0-tau]) Following Oral Administration of Ezogabine/Retigabine
Description: The steady state pharmacokinetic profile following oral administration of ezogabine/retigabine included determining the area under the curve over the dosing interval (AUC[0-tau]). The area under the plasma concentration-time curve over the dosing interval (AUC[0-tau]) was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35 to estimate AUC(0-tau).
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35
Population: Pharmacokinetic Population: all participants in the All Subjects Population (defined as all participants who received at least one dose of study medication) for whom a pharmacokinetic sample was obtained and analyzed
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*Nanograms/Milliliter (h.ng/mL)
Groups:
- Regimen A: Ezogabine/Retigabine (E/R) 300 mg: Participants (par.) with a body weight of >50 kilograms (kg) received a starting dose of 300 milligrams per day (mg/day) ezogabine/retigabine adminstered as 100 mg immediate release (IR) tablets three times a day (TID) orally and underwent weekly up-titration at a frequency of no more than once per week. The TID dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
- Regimen A: E/R 300/450 mg Then 600 mg: Par. with a body weight of >50 kg received a starting dose of 300 mg/day ezogabine/retigabine administered as 100 mg IR tablets TID orally and underwent weekly up-titration at a frequency of no more than once per week. At week two (Day 14), par. received 450 mg/day administered as 150 mg IR tablets TID orally.At week 3 (Day 21), par. received 600 mg/day administered as 200 mg IR tablets TID orally. The TID dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
- Regimen A: E/R 300/450/ 600/750 mg Then 900 mg: Par. with a body weight of >50 kg received a starting dose of 300 mg/day ezogabine/retigabine administered as 100 mg IR tablets TID orally and underwent weekly up-titration at a frequency of no more than once per week. At week two (Day 14), par. received 450 mg/day administered as 150 mg IR tablets TID orally. At week 3 (Day 21), par. received 600 mg/day administered as 200 mg IR tablets TID orally. At week 4 (Day 28), par. received 750 mg/day administered as 250 mg IR tablets TID orally. At week 5 (Day 35), par. received 900 mg/day administered as 300 mg IR tablets TID orally. The TID daily dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
Hour*Nanograms/Milliliter (h.ng/mL) | 1680.0 [1162.4 to 2428.2] | 2558.8 [1873.4 to 3494.8] | 3783.8 [1059.6 to 13512.0]

2. Primary Outcome: Apparent Clearance (CL/F) Following Oral Administration of Ezogabine/Retigabine
Description: Clearance (CL/F) is defined as dose/AUC(0-tau). Blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35 to estimate CL/F.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35
Population: Pharmacokinetic Population
Measure: Geometric Mean (95% Confidence Interval); unit: Liters/Hour
Groups:
- Regimen A: Ezogabine/Retigabine (E/R) 300 mg: Participants with a body weight of >50 kilograms (kg) received a starting dose of 300 milligrams per day (mg/day) ezogabine/retigabine adminstered as 100 mg immediate release (IR) tablets three times a day (TID) orally and underwent weekly up-titration at a frequency of no more than once per week. The TID dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
Liters/Hour | 178.6 [123.5 to 258.1] | 234.5 [171.7 to 320.3] | 237.9 [66.6 to 849.4]

3. Primary Outcome: Maximum Observed Concentration (Cmax) and Pre-dose (Trough) Concentration at the End of the Dosing Interval (Ctau) Following Oral Administration of Ezogabine/Retigabine
Description: Cmax is defined as the first occurrence of the maximum observed plasma concentration. Ctau refers to the pre-dose (trough) concentration after the dosing interval which is equal to the minimum observed concentration (Cmin) at Steady State. Blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35 to estimate Cmax and Ctau.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35
Population: Pharmacokinetic Population
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms/Milliliter (ng/mL)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
Nanograms/Milliliter (ng/mL)
  Cmax | 370.0 [260.9 to 524.7] | 535.9 [344.4 to 833.8] | 750.9 [289.8 to 1945.3]
  Ctau | 105.32 [58.70 to 188.98] | 199.77 [140.67 to 283.72] | 287.48 [44.38 to 1862.12]

4. Primary Outcome: Apparent Volume of Distribution (Vd/F) Following Oral Administration of Ezogabine/Retigabine
Description: The volume of distribution (Vd/F) is defined as MRT*CL/F, where MRT is the mean residence time (calculated as AUMC[0-tau]/AUC[0-tau], where AUMC[0-tau] is the area under the first moment curve determined as the area under the concentration*time versus time curve). Blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35 to estimate the apparent volume of distribution.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35
Population: Pharmacokinetic Population. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 3 | 3 | 1
Liters | 1130.9 [511.1 to 2502.1] | 2118.0 [539.4 to 8315.8] | 1934.3 [NA to NA] — Although 3 subjects were on this dose level during the study, only 1 provided data to calculate Volume of Distribution therefore the 95% CI is not available because of small sample size (n=1).

5. Secondary Outcome: Number of Participants With Any Adverse Event (AE)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Time Frame: From the start of the first titration until follow-up (assessed up to 46 days)
Population: All Subjects Population: all participants who received at least one dose of study medication
Measure: Number; unit: Participants
Groups:
- Regimen A: Ezogabine/Retigabine 300 mg: Participants with a body weight of >50 kg received a starting dose of 300 mg/day ezogabine/retigabine administerd as 100 mg IR tablets TID orally and underwent weekly up-titration at a frequency of no more than once per week. The TID dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
- Regimen A: Ezogabine/Retigabine 300 mg, Then 450 mg: Participants with a body weight of >50 kg received a starting dose of 300 mg/day ezogabine/retigabine administered as 100 mg IR tablets TID orally and underwent weekly up-titration at a frequency of no more than once per week. These participants then received an uptitrated dose of 450 mg/day ezogabine/retigabine as 150 mg IR tablets TID orally. The TID daily dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
- Regimen A: Ezogabine/Retigabine 300/450 mg, Then 600 mg: Participants with a body weight of >50 kg received a starting dose of 300 mg/day ezogabine/retigabine administered as 100 mg IR tablets TID orally and underwent weekly up-titration at a frequency of no more than once per week. These participants received an up-titrated dose of 450 mg/day ezogabine/retigabine (as 150 mg IR tablets TID orally) initially, then received an up-titrated dose of 600 mg/day ezogabine/retigabine as 200 mg IR tablets TID orally. The TID daily dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
- Regimen A: Ezogabine/Retigabine 300/450/600 mg, Then 750 mg: Participants with a body weight of >50 kg received a starting dose of 300 mg/day ezogabine/retigabine as 100 mg IR tablets TID orally and underwent weekly up-titration at a frequency of no more than once per week. These participants received up-titrated doses of ezogabine/retigabine 450 mg and 600 mg (as 150 mg IR and 200 mg IR tablets, respectively, TID orally) initially, then received an up-titrated dose of 750 mg/day ezogabine/retigabine as 250 mg IR tablets TID orally. The TID daily dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
- Regimen A: Ezogabine/Retigabine 300/450/600/750, Then 900 mg: Participants with a body weight of >50 kg received a starting dose of 300 mg/day ezogabine/retigabine as 100 mg IR tablets TID orally and underwent weekly up-titration at a frequency of no more than once per week. These participants received up-titrated doses of ezogabine/retigabine 450 mg, 600 mg, and 750 mg (as 150 mg IR, 200 mg IR, and 250 mg IR tablets, respectively, TID orally) initially, then received an up-titrated dose of 900 mg/day ezogabine/retigabine as 300 mg IR tablets TID orally. The TID daily dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
Arm/Group | Regimen A: Ezogabine/Retigabine 300 mg | Regimen A: Ezogabine/Retigabine 300 mg, Then 450 mg | Regimen A: Ezogabine/Retigabine 300/450 mg, Then 600 mg | Regimen A: Ezogabine/Retigabine 300/450/600 mg, Then 750 mg | Regimen A: Ezogabine/Retigabine 300/450/600/750, Then 900 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 3
Participants | 1 | 1 | 1 | 0 | 0

6. Secondary Outcome: Change From Baseline in Albumin and Total Protein at Day 7 Post Each Up-titration
Description: Change from baseline was calculated 7 days after each up-titration (Day 7 for 300 mg/day dose; Day 21 for up-titration to 600 mg/day dose; Day 35 for up-titration to 900 mg/day dose) by subtracting the baseline value from the individual post-dose values. Baseline is defined as the Screening visit.
Time Frame: Baseline (Screening), Day 7, Day 21, and Day 35
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: Grams per Liter (G/L)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
Grams per Liter (G/L)
  Albumin, n=4, 4, 3 | -3.8 (0.96) | -3.0 (3.46) | -0.7 (3.06)
  Total protein, n=4, 4, 3 | -4.0 (2.94) | -3.5 (3.79) | -0.7 (5.03)

7. Secondary Outcome: Change From Baseline in Alkaline Phosphatase, Alanine Amino Transferase, Aspartate Amino Transferase, and Gamma Glutamyl Transferase at Day 7 Post Each Up-titration
Description: as for outcome 6
Time Frame: Baseline (Screening), Day 7, Day 21, and Day 35
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: International Units per Liter (IU/L)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
International Units per Liter (IU/L)
  Alkaline phosphatse, n=4, 4, 3 | -5.8 (16.17) | 10.3 (35.93) | 5.0 (6.93)
  Alanine amino transferase, n=4, 4, 3 | -2.0 (2.16) | 35.0 (74.02) | -1.0 (2.00)
  Aspartate amino transferase, n=4, 4, 3 | -0.8 (2.50) | 10.8 (17.75) | 1.7 (3.21)
  Gamma glutamyl transferase, n=3, 3, 2 | -1.3 (0.58) | 111.0 (181.06) | 50.5 (47.38)

8. Secondary Outcome: Change From Baseline in Direct Bilirubin, Total Bilirubin, Creatinine, and Uric Acid at Day 7 Post Each Up-titration
Description: as for outcome 6
Time Frame: Baseline (Screening), Day 7, Day 21, and Day 35
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Micromoles per liter (UMOL/L)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
Micromoles per liter (UMOL/L)
  Direct bilirubin, n=1, 2, 1 | 2.7360 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | 2.7360 (3.86929) | -0.8550 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point.
  Total bilirubin, n=4, 4, 3 | 0.855 (2.2076) | 2.138 (2.5650) | 4.560 (0.9873)
  Creatinine, n=4, 4, 3 | 1.3260 (1.14124) | -4.1990 (5.02015) | 0.5893 (3.34677)
  Uric acid, n=4, 3, 1 | 16.3570 (19.04289) | 15.8613 (36.34288) | 23.7920 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point.

9. Secondary Outcome: Change From Baseline in Calcium, Chloride, Carbon Dioxide Content/Bicarbonate, Glucose, Potassium, Sodium, Inorganic Phosphorus, and Urea/Blood Urea Nitrogen (BUN) at Day 7 Post Each Up-titration
Description: as for outcome 6
Time Frame: Baseline (Screening), Day 7, Day 21, and Day 35
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimoles per liter (MMOL/L)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
Millimoles per liter (MMOL/L)
  Calcium, n=4, 4, 3 | 0.00624 (0.062375) | -0.04366 (0.117689) | 0.02495 (0.194866)
  Chloride, n=4, 4, 3 | 1.8 (0.96) | 3.0 (0.82) | 3.0 (1.73)
  Carbon dioxide content/bicarbonate, n=4, 4, 3 | 0.8 (3.50) | -1.5 (1.73) | -2.7 (2.08)
  Glucose, n=4, 4, 3 | 0.69388 (1.184069) | 0.15265 (0.821317) | 0.29605 (0.279394)
  Potassium, n=4, 4, 3 | 0.08 (0.206) | 0.17 (0.574) | 0.20 (0.624)
  Sodium, n=4, 4, 3 | 1.8 (0.50) | 2.0 (1.83) | 2.3 (3.06)
  Inorganic phosphorus, n=4, 3, 1 | -0.39555 (0.727481) | -0.04305 (0.189202) | 0.09687 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point.
  Urea/BUN, n=4, 4, 3 | -0.3570 (1.23668) | 0.7140 (0.71400) | 1.3090 (0.74315)

10. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils (Total ANC [Total Absolute Neutrophil Count]), Platelet Count, and White Blood Cell Count at Day 7 Post Each Up-titration
Description: as for outcome 6
Time Frame: Baseline (Screening), Day 7, Day 21, and Day 35
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Giga (10^9) cells per liter (GI/L)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
Giga (10^9) cells per liter (GI/L)
  Basophils, n=3, 3, 2 | 0.03 (0.062) | 0.04 (0.053) | 0.00 (0.006)
  Eosinophils, n=3, 3, 2 | 0.07 (0.059) | 0.09 (0.200) | 0.10 (0.005)
  Lymphocytes, n=3, 3, 2 | 14.77 (26.358) | -0.45 (0.654) | -0.65 (0.918)
  Monocytes, n=3, 3, 2 | -0.04 (0.347) | 0.09 (0.101) | 0.05 (0.065)
  Total neutrophils, n=3, 3, 2 | 14.90 (24.176) | -0.11 (0.370) | 0.61 (0.263)
  Platelet count, n=4, 4, 3 | -17.0 (40.12) | -15.8 (34.32) | -1.3 (17.16)
  White blood cell count, n=4, 4, 3 | 0.393 (1.2125) | -0.600 (0.6272) | -0.583 (1.3345)

11. Secondary Outcome: Change From Baseline in Hemoglobin and Mean Corpuscle Hemoglobin Concentration at Day 7 Post Each Up-titration
Description: as for outcome 6
Time Frame: Baseline (Screening), Day 7, Day 21, and Day 35
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
Grams per liter (G/L)
  Hemoglobin, n=4, 4, 3 | -3.0 (4.90) | -10.3 (6.85) | -2.0 (4.36)
  Mean corpuscle hemoglobin concentration, n=4, 4, 3 | -2.5 (2.38) | 0.3 (10.59) | -6.7 (4.93)

12. Secondary Outcome: Change From Baseline in Hematocrit at Day 7 Post Each Up-titration
Description: Change from baseline was calculated 7 days after each up-titration (Day 7 for 300 mg/day dose; Day 21 for up-titration to 600 mg/day dose; Day 35 for up-titration to 900 mg/day dose) by subtracting the baseline value from the individual post-dose values. Baseline is defined as the Screening visit. The International System of Units (SI) "Fraction of one unit (1)" is reported here.
Time Frame: Baseline (Screening), Day 7, Day 21, and Day 35
Population: All Subjects Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Fraction of one unit (1)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 4 | 4 | 3
Fraction of one unit (1) | -0.0057 (0.01452) | -0.0303 (0.02198) | 0.0017 (0.1201)

13. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin at Day 7 Post Each Up-titration
Description: as for outcome 6
Time Frame: Baseline (Screening), Day 7, Day 21, and Day 35
Population: All Subjects Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms (PG) per cell (PG/cell)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 4 | 4 | 3
Picograms (PG) per cell (PG/cell) | -0.07 (0.126) | 0.15 (0.569) | -0.23 (0.153)

14. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume at Day 7 Post Each Up-titration
Description: as for outcome 6
Time Frame: Baseline (Screening), Day 7, Day 21, and Day 35
Population: All Subjects Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters (FL)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 4 | 4 | 3
Femtoliters (FL) | 0.52 (1.056) | 0.45 (1.034) | 1.00 (1.000)

15. Secondary Outcome: Change From Baseline in Red Blood Cell Count at Day 7 Post Each Up-titration
Description: as for outcome 6
Time Frame: Baseline (Screening), Day 7, Day 21, and Day 35
Population: All Subjects Population. Only those participants available at the specified time point were analyzed.
Measure: Mean (Standard Deviation); unit: 10^12 cells/L (TI/L)
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 4 | 4 | 3
10^12 cells/L (TI/L) | -0.090 (0.1463) | -0.357 (0.2304) | -0.030 (0.1136)

16. Secondary Outcome: Number of Participants With the Indicated Urinalysis Parameter Dipstick Test Results From Screening to Follow-up
Description: Urinalysis parameters analyzed included: urine occult blood (UOB), urine glucose (UG), urine ketones (UK), and urine protein (UP). The dipstick was a strip used to detect the presence or absence of these parameters in the urine sample. The dipstick test provides results in a semi-quantitative manner, and results can be read as negative (Neg), Trace, and 80, indicating proportional concentrations in the urine sample. Urinalysis parameters were assessed at Titration 1 (T1; 300 mg/day), Titration 2 (T2; 450 mg/day), Titration 3 (T3; 600 mg/day), Titration 4 (T4; 750 mg/day), and Titration 5 (T5; 900 mg/day).
Time Frame: Screening, Day 1 (D1), Day 7 (D7), Day 14 (D14), Day 21 (D21), Day 28 (D28), Day 35 (D35), and at the Follow-up Visit (up to Day 46)
Population: All Subjects Population (ASP). Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X in the category titles). Different participants may have been analyzed at different time points and for different parameters, so the overall number of participants analyzed reflects everyone in the ASP.
Measure: Number; unit: Participants
Groups:
- Regimen A: Ezogabine/Retigabine 300 mg, Then 450 mg: Participants with a body weight of >50 kg received a starting dose of 300 mg/day ezogabine/retigabine administered as 100 mg IR tablets TID orally and underwent weekly up-titration at a frequency of no more than once per week. These participants then received an up-titrated dose of 450 mg/day ezogabine/retigabine as 150 mg IR tablets TID orally. The TID daily dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
- Regimen A: Ezogabine/Retigabine 300/450/600 mg, Then 750 mg: Participants with a body weight of>50 kg received a starting dose of 300 mg/day ezogabine/retigabine as 100 mg IR tablets TID orally and underwent weekly up-titration at a frequency of no more than once per week. These participants received up-titrated doses of ezogabine/retigabine 450 mg and 600 mg (as 150 mg IR and 200 mg IR tablets, respectively, TID orally) initially, then received an up-titrated dose of 750 mg/day ezogabine/retigabine as 250 mg IR tablets TID orally. The TID daily dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
Arm/Group | Regimen A: Ezogabine/Retigabine 300 mg | Regimen A: Ezogabine/Retigabine 300 mg, Then 450 mg | Regimen A: Ezogabine/Retigabine 300/450 mg, Then 600 mg | Regimen A: Ezogabine/Retigabine 300/450/600 mg, Then 750 mg | Regimen A: Ezogabine/Retigabine 300/450/600/750, Then 900 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 3
Participants
  UOB, T1, D1, 80, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UOB, T1, D1, Negative, n=5, 0, 0, 0, 0 | 4 | 0 | 0 | 0 | 0
  UOB, T1, D1, Trace, n=5, 0, 0, 0, 0 | 1 | 0 | 0 | 0 | 0
  UOB, T1, D7, 80, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UOB, T1, D7, Negative, n=5, 0, 0, 0, 0 | 4 | 0 | 0 | 0 | 0
  UOB, T1, D7, Trace, n=5, 0, 0, 0, 0 | 1 | 0 | 0 | 0 | 0
  UOB, T2, D7, 80, n=0, 5, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UOB, T2, D7, Negative, n=0, 5, 0, 0, 0 | 0 | 5 | 0 | 0 | 0
  UOB, T2, D7, Trace, n=0, 5, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UOB, T3, D7, 80, n=0, 0, 4, 0, 0 | 0 | 0 | 0 | 0 | 0
  UOB, T3, D7, Negative, n=0, 0, 4, 0, 0 | 0 | 0 | 3 | 0 | 0
  UOB, T3, D7, Trace, n=0, 0, 4, 0, 0 | 0 | 0 | 1 | 0 | 0
  UOB, T3, D14, 80, n=0, 0, 1, 0, 0 | 0 | 0 | 0 | 0 | 0
  UOB, T3,D14, Negative, n=0, 0, 1, 0, 0 | 0 | 0 | 1 | 0 | 0
  UOB, T3, D14, Trace, n=0, 0, 1, 0, 0 | 0 | 0 | 0 | 0 | 0
  Urine Occult Blood, T4, D7, 80, n=0,0,0,3,0 | 0 | 0 | 0 | 0 | 0
  UOB, T4, D7, Negative, n=0, 0, 0, 3, 0 | 0 | 0 | 3 | 0 | 0
  Urine Occult Blood, T4, D7, Trace, n=0,0,0,3,0 | 0 | 0 | 0 | 0 | 0
  UOB, T5, D7, 80, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 0
  UOB, T5, D7, Negative, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 2
  UOB, T5, D7, Trace, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 1
  UG, T1, D1, 80, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UG, T1, D1, Negative, n=5, 0, 0, 0, 0 | 5 | 0 | 0 | 0 | 0
  UG, T1, D1, Trace, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UG, T1, D7, 80, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UG, T1, D7, Negative, n=5, 0, 0, 0, 0 | 5 | 0 | 0 | 0 | 0
  UG, T1, D7, Trace, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UG, T2, D7, 80, n=0, 5, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UG, T2, D7, Negative, n=0, 5, 0, 0, 0 | 0 | 5 | 0 | 0 | 0
  UG, T2, D7, Trace, n=0, 5, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UG, T3, D7, 80, n=0, 0, 4, 0, 0 | 0 | 0 | 0 | 0 | 0
  UG, T3, D7, Negative, n=0, 0, 4, 0, 0 | 0 | 0 | 4 | 0 | 0
  UG, T3, D7, Trace, n=0, 0, 4, 0, 0 | 0 | 0 | 0 | 0 | 0
  UG, T3, D14, 80, n=0, 0,1,0,0 | 0 | 0 | 0 | 0 | 0
  UG, T3, D14, Negative, n=0, 0, 1, 0, 0 | 0 | 0 | 1 | 0 | 0
  UG, T3, D14, Trace, n=0, 0, 1, 0, 0 | 0 | 0 | 0 | 0 | 0
  UG, T4, D7, 80, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 0 | 0
  UG, T4, D7, Negative, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 4 | 0
  UG, T4, D7, Trace, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 0 | 0
  UG, T5, D7, 80, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 0
  UG, T5, D7, Negative, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 3
  UG, T5, D7, Trace, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 0
  UK, T1, D1, 80, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UK, T1, D1, Negative, n=5, 0, 0, 0, 0 | 5 | 0 | 0 | 0 | 0
  UK, T1, D1, Trace, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UK, T1, D7, 80, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UK, T1, D7, Negative, n=5, 0, 0, 0, 0 | 5 | 0 | 0 | 0 | 0
  UK, T1, D7, Trace, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UK, T2, D7, 80, n=0, 5, 0, 0, 0 | 0 | 1 | 0 | 0 | 0
  UK, T2, D7, Negative, n=0, 5, 0, 0, 0 | 0 | 3 | 0 | 0 | 0
  UK, T2, D7, Trace, n=0, 5, 0, 0, 0 | 0 | 1 | 0 | 0 | 0
  UK, T3, D7, 80, n=0, 0, 4, 0, 0 | 0 | 0 | 0 | 0 | 0
  UK, T3, D7, Negative, n=0, 0, 4, 0, 0 | 0 | 0 | 4 | 0 | 0
  UK, T3, D7, Trace, n=0, 0, 4, 0, 0 | 0 | 0 | 0 | 0 | 0
  UK, T3, D14, 80, n=0, 0, 1, 0, 0 | 0 | 0 | 0 | 0 | 0
  UK, T3, D14, Negative, n=0, 0, 1, 0, 0 | 0 | 0 | 1 | 0 | 0
  UK, T3, D14, Trace, n=0, 0, 1, 0, 0 | 0 | 0 | 0 | 0 | 0
  UK, T4, D7, 80, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 0 | 0
  UK, T4, D7, Negative, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 4 | 0
  UK, T4, D7, Trace, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 0 | 0
  UK, T5, D7, 80, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 0
  UK, T5, D7, Negative, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 3
  UK, T5, D7, Trace, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 0
  UP, T1, D1, 80, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UP, T1, D1, Negative, n=5, 0, 0, 0, 0 | 4 | 0 | 0 | 0 | 0
  UP, T1, D1, Trace, n=5, 0, 0, 0, 0 | 1 | 0 | 0 | 0 | 0
  UP, T1, D7, 80, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UP, T1, D7, Negative, n=5, 0, 0, 0, 0 | 5 | 0 | 0 | 0 | 0
  UP, T1, D7, Trace, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UP, T2, D7, 80, n=0, 5, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  UP, T2, D7, Negative, n=0, 5, 0, 0, 0 | 0 | 4 | 0 | 0 | 0
  UP, T2, D7, Trace, n=0, 5, 0, 0, 0 | 0 | 1 | 0 | 0 | 0
  UP, T3, D7, 80, n=0, 0, 4, 0,0 | 0 | 0 | 0 | 0 | 0
  UP, T3, D7, Negative, n=0, 0, 4, 0, 0 | 0 | 0 | 3 | 0 | 0
  UP, T3, D7, Trace, n=0, 0, 4, 0, 0 | 0 | 0 | 1 | 0 | 0
  UP, T3, D14, 80, n=0, 0, 1, 0, 0 | 0 | 0 | 0 | 0 | 0
  UP, T3, D14, Negative, n=0, 0, 1, 0, 0 | 0 | 0 | 1 | 0 | 0
  UP, T3, D14, Trace, n=0, 0, 1, 0, 0 | 0 | 0 | 0 | 0 | 0
  UP, T4, D7, 80, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 0 | 0
  UP, T4, D7, Negative, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 4 | 0
  UP, T4, D7, Trace, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 0 | 0
  UP, T5, D7, 80, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 0
  UP, T5, D7, Negative, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 3
  UP, T5, D7, Trace, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Percent Change From Baseline in 28-day Seizure Frequency Rate
Description: Participants or their caregivers recorded the number of seizures experienced by the participant, by seizure type (e.g., simple partial seizure [seizure that affects only a small region of the brain; consciousness is unaffected], complex partial seizure [seizure associated with unilateral cerebral hemisphere involvement and causing impairment of awareness or responsiveness], etc.), as well as by duration of episodes of innumerable seizure activity, in their daily diaries during all phases of this study. Percent change from baseline is defined as 100 * (rate in a given period minus the baseline rate) / (baseline rate). baseline seizures are defined as those seizures that occurred after Screening and before the start of the treatment. Post-baseline seizures are defined as those seizures that occurred from the start of the treatment until the start of Follow-up. Seizure frequency rate was computed as: 28 * (number of seizures during given period / number of days in given period).
Time Frame: Baseline (Screening) and until Follow-up or early discontinuation (assessed up to 46 days)
Population: All Subjects Population. Only participants with baseline and post-baseline seizure measurements were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Regimen A: Ezogabine/Retigabine 300/450/600/750, Then 900 mg: Participants recieved an initial dose of ezogabine/retigabine 300 mg/day administered as 100 mg IR tablets TID orally and underwent weekly up-titration at Weeks 1, 3, and 5. Dose titration occurred no more than once per week, with participants receiving up-titrated daily doses of 450 mg (150 mg TID), 600 mg (200 mg TID), 750 mg (250 mg TID), and 900 mg (300 mg TID) at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
Arm/Group | Regimen A: Ezogabine/Retigabine 300/450/600/750, Then 900 mg
Number analyzed (Participants) | 5
Percent change | -41.5 (29.95)

18. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero (Pre-dose) to the Last Time of Quantifiable Concentration (AUC [0-t]) for the N-acetyl Metabolite of Ezogabine/Retigabine
Description: The area under the curve was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations. Blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35 to assess the plasma n-acetyl metabolite (NAMR) of ezogabine/retigabine following oral administration of ezogabine/retigabine.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
h*ng/mL | 2222.1 [1531.4 to 3224.4] | 3479.2 [2374.0 to 5099.0] | 5000.6 [1528.9 to 16355.7]

19. Secondary Outcome: Pre-dose (Trough) Concentration at the End of the Dosing Interval (Ctau) for the N-acetyl Metabolite of Ezogabine/Retigabine
Description: Ctau refers to the pre-dose (trough) concentration at the end of the dosing interval which is equivalent to the minimum observed concetration (Cmin) at Steady State. Blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35 to assess the Ctau for n-acetyl metabolite (NAMR) of ezogabine/retigabine following oral administration of ezogabine/retigabine.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Regimen A: Ezogabine/Retigabine (E/R) 300 mg: Participants with a body weight of >50 kilograms (kg) received a starting dose of 300 milligrams per day (mg/day) ezogabine/retigabine adminstered as 100 mg immediate release (IR) tablets three times a day (TID) orally and underwent weekly upitration at a frequency of no more than once per week. The TID dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
ng/mL | 170.51 (86.32) [86.32 to 336.82] | 307.85 [190.25 to 498.14] | 415.66 [120.74 to 1430.93]

20. Secondary Outcome: Time to Maximum Concentration (Tmax) Following Oral Administration of Ezogabine/Retigabine
Description: Blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35 to assess plasma Tmax.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35
Population: PK Population
Measure: Median (Full Range); unit: Hours
Groups:
- Regimen A: Ezogabine/Retigabine (E/R)300 mg: Participants with a body weight of >50 kilograms (kg) received a starting dose of 300 milligrams per day (mg/day) ezogabine/retigabine adminstered as 100 mg immediate release (IR) tablets three times a day (TID) orally and underwent weekly up-titration at a frequency of no more than once per week. The TID dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
- Regimen A: E/R 300/450/ 600/750 Then 900 mg: Par. with a body weight of >50 kg received a starting dose of 300 mg/day ezogabine/retigabine administered as 100 mg IR tablets TID orally and underwent weekly up-titration at a frequency of no more than once per week. At week two (Day 14), par. received 450 mg/day administered as 150 mg IR tablets TID orally. At week 3 (Day 21), par. received 600 mg/day administered as 200 mg IR tablets TID orally. At week 4 (Day 28), par. received 750 mg/day administered as 250 mg IR tablets TID orally. At week 5 (Day 35), par. received 900 mg/day administered as 300 mg IR tablets TID orally. The TID daily dosing regimen was administered at an 8-hour dosing interval or a 6-, 6-, 12-hour dosing interval.
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R)300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 Then 900 mg
Number analyzed (Participants) | 5 | 4 | 3
Hours | 1.000 [0.50 to 1.08] | 1.550 [0.50 to 8.00] | 2.000 [0.50 to 6.00]

21. Secondary Outcome: Plasma Half Life at Steady State (t1/2) Following Oral Administration of Ezogabine/Retigabine
Description: Blood samples were collected at pre-dose and at 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35 to assess plasma t1/2. Steady-state t1/2 is derived as (Vd/F) / (CL/F), where Vd/F is defined as the apparent volume of distribution after extravascular (e.g., oral) administration, and CL/F is defined as the apparent clearance following oral dosing.
Time Frame: Pre-dose and 0.5, 1, 1.5, 2, 4, 6, and 8 hours post-dose on Day 7, Day 21, and Day 35
Population: PK Population. Only those participants available at the indicated time point were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | Regimen A: Ezogabine/Retigabine (E/R) 300 mg | Regimen A: E/R 300/450 mg Then 600 mg | Regimen A: E/R 300/450/ 600/750 mg Then 900 mg
Number analyzed (Participants) | 3 | 3 | 1
Hours | 4.168 [2.363 to 7.350] | 5.897 [0.962 to 36.160] | 3.473 [NA to NA] — The 95% CI cannot be calculated because only one participant has been analyzed in this treatment arm at this time point

22. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: An ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT interval corrected for heart rate (QTc intervals) was used. Measurements were taken 7 days after each up-titration (Day 7 for 300 mg/day dose; Day 14 for up-titration to 450 mg/day dose; Day 21 for up-titration to 600 mg/day dose; Day 28 for up-titration to 750 mg/day dose; Day 35 for up-titration to 900 mg/day dose). ECG parameters were assessed at Titration 1 (T1; 300 mg/day): Day 1 pre-dose, Day 1 at 3 hours (h), pre-dose, and 3 h post-dose. Titration 2 (T2; 450 mg/day): Day 7. Titration 3 (T3; 600 mg/day): pre-dose and 3 h post-dose. Titration 3 Dose Held (T3DH): pre-dose. Titration 4 (T4; 750 mg/day): Day 7. Titration 5 (T5; 900 mg/day): pre-dose and 3 h post-dose. The number of participants with abnormal (Abn) clinically significant (CS) and not clinically significant (NCS) ECG findings was recorded. The investigator determined if an ECG finding was CS or NCS.
Time Frame: Baseline (Screening) and Day 7 post up-titration, up to Day 35
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X, X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Number; unit: Participants
Arm/Group | Regimen A: Ezogabine/Retigabine 300 mg | Regimen A: Ezogabine/Retigabine 300 mg, Then 450 mg | Regimen A: Ezogabine/Retigabine 300/450 mg, Then 600 mg | Regimen A: Ezogabine/Retigabine 300/450/600 mg, Then 750 mg | Regimen A: Ezogabine/Retigabine 300/450/600/750, Then 900 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 3
Participants
  T1, Day 1 pre-dose, Abn NCS, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  T1, Day 1 pre-dose, Abn CS, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  T1, Day 1, 3 h, Abn NCS, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  T1, Day 1, 3 h, Abn CS, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  T1, pre-dose, Abn NCS, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  T1, pre-dose, Abn CS, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  T1, 3 h, Abn NCS, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  T1, 3 h, Abn CS, n=5, 0, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  T2, Day 7, Abn NCS, n=0, 5, 0, 0, 0 | 0 | 1 | 0 | 0 | 1
  T2, Day 7, Abn CS, n=0, 5, 0, 0, 0 | 0 | 0 | 0 | 0 | 0
  T3, pre-dose, Abn NCS, n=0, 0, 4, 0, 0 | 0 | 0 | 0 | 0 | 0
  T3, pre-dose, Abn CS, n=0, 0, 4, 0, 0 | 0 | 0 | 0 | 0 | 0
  T3, 3 h, Abn NCS, n=0, 0, 4, 0, 0 | 0 | 0 | 0 | 0 | 0
  T3, 3 h, Abn CS, n=0, 0, 4, 0, 0 | 0 | 0 | 0 | 0 | 0
  T3DH, pre-dose, Abn NCS, n=0, 0, 1, 0, 0 | 0 | 0 | 0 | 0 | 0
  T3DH, pre-dose, Abn CS, n=0, 0, 1, 0, 0 | 0 | 0 | 0 | 0 | 0
  T4, Day 7, Abn NCS, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 0 | 0
  T4, Day 7, Abn CS, n=0, 0, 0, 4, 0 | 0 | 0 | 0 | 0 | 0
  T5, pre-dose, Abn NCS, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 1
  T5, pre-dose, Abn CS, n=0, 0, 0, 0, 3 | 0 | 0 | 0 | 0 | 0
  T5, 3 h, Abn NCS, n=0, 0, 0, 0, 2 | 0 | 0 | 0 | 0 | 0
  T5, 3 h, Abn CS, n=0, 0, 0, 0, 2 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points
Description: Vital sign assessment included the measurement of systolic and diastolic blood pressure at Titration 1 (T1; 300 mg/day): Day 1 pre-dose, Day 1 at 3 hours (h), Day 7 pre-dose, and 3 h post dose. Titration 2 (T2; 450 mg/day): Day 7. Titration 3 (T3; 600 mg/day): Day 21 pre-dose and 3 h post-dose. Titration 3 Dose Held (T3DH): pre-dose. Titration 4 (T4; 750 mg/day): Day 7. Titration 5 (T5; 900 mg/day): Day 35 pre-dose and 3 h post-dose. Measurements were taken 7 days after each up-titration (Day 7 for 300 mg/day dose; Day 14 for up-titration to 450 mg/day dose; Day 21 for up-titration to 600 mg/day dose; Day 28 for up-titration to 750 mg/day dose; Day 35 for up-titration to 900 mg/day dose). Change from baseline was calculated by subtracting the baseline value from the individual post-dose values. Baseline is defined as as the Day 1 pre-dose value.
Time Frame: Baseline (Screening) and Day 7 post up-titration, up to Day 35
Population: All Subjects Population. Only those par. available at the specified time points were analyzed(represented by n=X, X, X, X, X in the category titles). Different par. may have been analyzed at different time points and for different parameters, so the overall number of par. analyzed reflects everyone in the All Subjects Population.
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Regimen A: Ezogabine/Retigabine 300 mg | Regimen A: Ezogabine/Retigabine 300 mg, Then 450 mg | Regimen A: Ezogabine/Retigabine 300/450 mg, Then 600 mg | Regimen A: Ezogabine/Retigabine 300/450/600 mg, Then 750 mg | Regimen A: Ezogabine/Retigabine 300/450/600/750, Then 900 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 3
Millimeters of Mercury (mmHg)
  SBP, T1, Day 1 3h, n=5, 0, 0, 0, 0 | 2.8 (6.02) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  SBP, T1, Day 7 Pre-dose, n=5, 0, 0, 0, 0 | 2.6 (5.18) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  SBP, T1, Day 7 3h, n=5, 0, 0, 0, 0 | -1.2 (8.81) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  SBP, T2, Day 7, n=0, 5, 0, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 5.4 (4.39) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  SBP, T3, Day 21 Pre-dose, n=0, 0, 4, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 11.3 (11.62) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  SBP, T3, Day 21 3h, n=0, 0, 4, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 3.0 (10.68) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  SBP, T3DH, Pre-dose, n=0, 0, 1, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 13.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  SBP, T4, Day 28, n=0, 0, 0, 4, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 3.0 (3.27) | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  SBP, T5, Day 35 Pre-dose, n=0, 0, 0, 0, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 8.7 (13.32)
  SBP, T5, Day 35 3h, n=0, 0, 0, 0, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 5.3 (10.97)
  DBP, T1, Day 1 3h, n=5, 0, 0, 0, 0 | 1.4 (7.92) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  DBP, T1, Pre-dose, n=5, 0, 0, 0, 0 | 0.2 (4.60) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  DBP, T1, 3h, n=5, 0, 0, 0, 0 | 4.4 (5.81) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  DBP, T2, Day 7, n=0, 5, 0, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -0.2 (15.55) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  DBP, T3, Pre-dose, n=0, 0, 4, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 1.8 (4.65) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  DBP, T3, 3h, n=0, 0, 4, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 3.8 (12.89) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  DBP, T3DH, Pre-dose, n=0, 0, 1, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 23.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  DBP, T4, Day 7, n=0, 0, 0, 4, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | -0.3 (2.99) | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  DBP, T5, Pre-dose, n=0, 0, 0, 0, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 7.3 (12.70)
  DBP, T5, 3h, n=0, 0, 0, 0, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 3.7 (16.77)

24. Secondary Outcome: Change From Baseline in Heart Rate (HR)
Description: Vital sign assessment included heart rate measurement and was assessed at Titration 1 (T1; 300 mg/day): Day 1 pre-dose, Day 1 at 3 hours (h), pre-dose and 3 h post-dose. Titration 2 (T2; 450 mg/day): Day 7. Titration 3 (T3; 600 mg/day): pre-dose and 3 h post-dose. Titration 3 Dose Held (T3DH): pre-dose. Titration 4 (T4; 750 mg/day): Day 7. Titration 5 (T5; 900 mg/day): pre-dose and 3 h post-dose. Measurements were taken 7 days after each up-titration (Day 7 for 300 mg/day dose; Day 14 for up-titration to 450 mg/day dose; Day 21 for up-titration to 600 mg/day dose; Day 28 for up-titration to 750 mg/day dose; Day 35 for up-titration to 900 mg/day dose). Change from baseline was calculated by subtracting the baseline value from the individual post-dose values. Baseline is defined as as the Day 1 pre-dose value.
Time Frame: Baseline (Screening) and Day 7 post up-titration, up to Day 35
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Beats per Minute (BPM)
Arm/Group | Regimen A: Ezogabine/Retigabine 300 mg | Regimen A: Ezogabine/Retigabine 300 mg, Then 450 mg | Regimen A: Ezogabine/Retigabine 300/450 mg, Then 600 mg | Regimen A: Ezogabine/Retigabine 300/450/600 mg, Then 750 mg | Regimen A: Ezogabine/Retigabine 300/450/600/750, Then 900 mg
Number analyzed (Participants) | 5 | 5 | 4 | 4 | 3
Beats per Minute (BPM)
  HR, T1, Day 1 3h, n=5, 0, 0, 0, 0 | 3.6 (11.26) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  HR, T1, Pre-dose, n=5, 0, 0, 0, 0 | -0.8 (7.22) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  HR, T1, 3h, n=5, 0, 0, 0, 0 | 2.8 (5.89) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  HR, T2, Day 7, n=0, 5, 0, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 8.2 (11.67) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  HR, T3, Pre-dose, n=0, 0, 4, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 0.5 (7.51) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  HR, T3, 3h, n=0, 0, 4, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 6.0 (5.48) | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  HR, T3DH, Pre-dose, n=0, 0, 1, 0, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 8.0 (NA) — The standard deviation cannot be calculated because only one participant has been analyzed in this treatment arm at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  HR, T4, Day 7, n=0, 0, 0, 4, 0 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 1.8 (6.18) | NA (NA) — No participants in this treatment arm were analyzed at this time point.
  HR, T5, Pre-dose, n=0, 0, 0, 0, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 1.7 (4.16)
  HR, T5, 3h, n=0, 0, 0, 0, 3 | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | NA (NA) — No participants in this treatment arm were analyzed at this time point. | 2.3 (4.16)

25. Secondary Outcome: Change From Baseline in Post Void Residual Ultrasound at Day 21
Description: A post void residual (PVR) bladder ultrasound was carried out as a measure of bladder function. PVR was clinically indicated following the occurrence of adverse events relating to the lower urinary tract (e.g., micturition difficulties, including urinary hesitancy or urinary retention). These assessments were also repeated following drug withdrawal following such events. A prompt follow-up PVR was recommended if a high score was obtained from a participant on the Pediatric Lower Urinary Tract Symptom scale (the PLUTS scale is a clinician-rated scale used to assess lower urinary tract symptoms, including urinary retention) and if the clinician felt that the participant was at risk or had symptoms of urinary retention. PVR was measured at Day 7 of Titration 3 (600 mg/day). Baseline is defined as the Screening visit.
Time Frame: Screening and Day 7 of Titration 3 (Day 21)
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: ML
Arm/Group | Regimen A: Ezogabine/Retigabine 300/450 mg, Then 600 mg
Number analyzed (Participants) | 4
ML | 14.4 (21.00)

26. Secondary Outcome: Number of Participants With the Indicated Neurological Abnormality
Description: Abnormal Central Nervous System (CNS) symptoms were assessed by a full and brief neurological examination. A full neurological examination included assessment of mental status, cranial nerves, gait, coordination, sensation, speech/language, muscle strength, muscle tone, and reflexes. A brief neurological examination included assessment of mental status, cranial nerves, gait, coordination, reflexes, and speech/language. Neurological parameters assessed were memory impairment, impaired intellect, decreased attention, psychomotor slowing, decreased muscle strength, hpertonia, somnolence, right and left bicpes, right and left brachioradialis, right and left knee, right and left ankle, and right and left planter response. Neurological examination was performed at Day 7 of Titration 3 (600 mg/day).
Time Frame: Screening and Day 7 of Titration 3 (Day 21)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Regimen A: Ezogabine/Retigabine 300/450 mg, Then 600 mg
Number analyzed (Participants) | 4
Participants
  Memory impairment | 0
  Impaired intellect | 0
  Decreased attention | 0
  Psychomotor slowing | 0
  Decreased muscle strength | 0
  Hypertonia | 0
  Somnolence | 1
  Bicep right | NA — Only a brief neurological exam was conducted therefore this value was not measured
  Bicep left | NA — Only a brief neurological exam was conducted therefore this value was not measured
  Brachioradialis right | NA — Only a brief neurological exam was conducted therefore this value was not measured
  Brachioradialis left | NA — Only a brief neurological exam was conducted therefore this value was not measured
  Knee right | NA — Only a brief neurological exam was conducted therefore this value was not measured
  Knee left | NA — Only a brief neurological exam was conducted therefore this value was not measured
  Ankle right | NA — Only a brief neurological exam was conducted therefore this value was not measured
  Ankle left | NA — Only a brief neurological exam was conducted therefore this value was not measured
  Planter response right | NA — Only a brief neurological exam was conducted therefore this value was not measured
  Planter response left | NA — Only a brief neurological exam was conducted therefore this value was not measured

ADVERSE EVENTS:
Time Frame: Adverse event data, volunteered by the participant, discovered by the investigator, or detected by other means, were collected from the start of study treatment until the Follow-up contact (maximum of 46 days).
Description: Serious adverse events (SAEs) and non-serious AEs were collected in members of the All Subjects Population, comprsised of all participants who received at least one dose of study medication.
Arm/Group | Regimen A: Ezogabine/Retigabine 300 mg | Regimen A: Ezogabine/Retigabine 300 mg, Then 450 mg | Regimen A: Ezogabine/Retigabine 300/450 mg, Then 600 mg | Regimen A: Ezogabine/Retigabine 300/450/600 mg, Then 750 mg | Regimen A: Ezogabine/Retigabine 300/450/600/750, Then 900 mg
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/4 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/5 | 1/5 | 1/4 | 0/4 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A: Ezogabine/Retigabine 300 mg (N=5) | Regimen A: Ezogabine/Retigabine 300 mg, Then 450 mg (N=5) | Regimen A: Ezogabine/Retigabine 300/450 mg, Then 600 mg (N=4) | Regimen A: Ezogabine/Retigabine 300/450/600 mg, Then 750 mg (N=4) | Regimen A: Ezogabine/Retigabine 300/450/600/750, Then 900 mg (N=3)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.